CLINICAL TRIAL: NCT05317169
Title: Aneurysm Genetic Risk in Patients With Changes in Quantitative Imaging Biomarkers Over Time
Brief Title: Aneurysm Genetic Risk in Patients With QIB Changes
Acronym: AnGen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Aichi Chien, PhD, Professor, University of California, Los Angeles
Other Study IDs: 16-001867
Record Dates: First submitted 2021-12-14; First posted 2022-04-07 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Brain Aneurysm
Keywords: Brain Aneurysm; Ruptured Brain Aneurysm; Aneurysm Growth; Brain Aneurysm Genetic Markers; Vascular Malformation
MeSH Terms: conditions — Intracranial Aneurysm; Vascular Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intracranial aneurysm rupture is a leading cause of hemorrhagic strokes which carry high mortality and disability rates as well as high healthcare costs. Unruptured intracranial aneurysms (UIA) are common in the general population, occurring in 1-2% of individuals. Previous studies have shown that UIA growth and rupture are strongly associated with each other, with growing aneurysms 9-12 times more likely to rupture, and nearly all aneurysms growing prior to rupture. Thanks to advanced medical imaging, UIA are now more and more often detected incidentally. However not all aneurysms qualify for preventive surgical or interventional procedures according to current International Study of Unruptured Intracranial Aneurysms (ISUIA) guidelines, and some must therefore be monitored for growth. Current guidelines are based heavily on size, an inconsistent predictor of future growth. To improve management strategies for individual patients and more comprehensively assess aneurysm risk, the investigators propose to identify risk factors related to growth.

Aneurysm etiology is multifactorial, with both genetic and environmental contributions to aneurysm formation, growth, and rupture. Exploring new risk factors based on aneurysm natural history and understanding the mechanisms underlying aneurysm rupture have been extensive research areas. As previous studies have shown that quantitative imaging biomarkers (QIB) can provide a more accurate assessment of the characteristics of aneurysms, the investigators propose a combined study which identifies QIB associated with aneurysm growth to identify factors related to growth.

DETAILED DESCRIPTION:
The objective of this study is to investigate intracranial aneurysms that have been followed with clinical 3D aneurysm images and create a matrix that can identify the risk of growth by integrating QIB with genetic predisposition risk factors. 120 Patients who have been followed by clinical aneurysm imaging study will be enrolled in this study. The study team will collect blood samples from the patients for genetic analysis.

To find the genetic factors, the blood samples will be processed with a focus on genetic variants 1) in pathways involved in endothelial and vascular function and 2) previously identified in genome-wide association studies of aneurysm risk. These analyses will include both common polymorphisms and rare alterations. These biomarkers have important implications for facilitating identification of high-risk subgroups for aneurysm growth and the development of improved evidence-based decision-making.

The investigators will perform aneurysm 3D analysis based on the aneurysm images to extract aneurysm QIB for these cases. Shape parameters such as aneurysm surface area shape indices will be collected for individual aneurysms as well as parameters capturing the aneurysm blood flow pattern. The study plans to address whether certain genetic variants for vascular function are present in patients with QIB change over time.

ELIGIBILITY:
Inclusion Criteria:

Patients with unruptured cerebral aneurysms followed yearly using non-invasive imaging techniques including Computed tomography (CT) and Magnetic resonance (MR) angiography.

Exclusion Criteria:

Patients with bleeding disorders. Patients who have severe intravenous CT or MR contrast allergy. Patients with evidence of kidney failure. Patients with severe claustrophobia. Patients with religious objections to phlebotomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UCLA patients who come for yearly CT or MR angiography for cerebral aneurysm surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2023-09-27 (Estimated); Study Completion 2023-09-27 (Estimated)

PRIMARY OUTCOMES:
Quantitative imaging biomarkers (QIB) change | 3 years
  Number of participants with changes in quantitative imaging biomarkers

SECONDARY OUTCOMES:
Genetic biomarkers in QIB change | 3 years
  Number of participants with genetic biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Aichi Chien, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States